CLINICAL TRIAL: NCT00212485
Title: Evaluation of the Role of Power Doppler Sonography in the Diagnosis of Hemophilic Joint Disease
Brief Title: Study to Evaluate the Use of Ultrasound in the Diagnosis of Hemophilic Joint Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Presbyterian Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Suchitra Acharya, MD, New York Presbyterian Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PDS
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Inherited Bleeding Disorders
Keywords: Hemophilia; Factor Deficiency; synovitis; sonogram
MeSH Terms: conditions — Hemophilia A; Synovitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Power Doppler Sonography — Power Doppler with gray-scale sonography is used to detect and quantify alterations in vascularity inside knee, elbow and ankle joints.
Procedure: MRI — Magnetic Resonance Imaging with intravenous gadolinium contrast will be done using a standardized protocol, including a spin echo T2 weighted image and gradient echo images.

SUMMARY:
The purpose of this study is to see whether power Doppler sonography (PDS) can be used to diagnose synovitis in patients with inherited bleeding disorders.

DETAILED DESCRIPTION:
Aim #1 - To determine if PDS can be used to diagnose synovial hypertrophy and inflammation in joint disease associated with inherited bleeding disorders. MRI will be used as a reference standard.

Aim #2 - To determine if PDS can be used to assess therapeutic response to treatment.

Aim #3 - To determine if PDS can be used as a screening tool for diagnosing early synovitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of inherited bleeding disorder

For Aim 1:

* Age of at least 6 years
* History of at least 4 bleeds in the same joint in the preceding 6 months
* Joint swelling, synovitis or deformity

For Aim 2:

* Meet inclusion criteria for Aim 1 and will be having a synovectomy

For Aim 3:

* Age of at least 1 year
* Have had at least 2 joint bleeds

Exclusion Criteria:

* Not meeting inclusion criteria

Ages: 1 Year to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 43 (Actual)
Dates: Start 2005-09; Primary Completion 2008-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Comparison of magnetic resonance imaging (MRI) and power Doppler sonograms on patients with target joint | Up to 1 month
Evaluation of PDS on patients with target joints pre and post synovectomy to assess response to therapeutic intervention | 1. day of synovectomy; 2. 6 months post synovectomy.
Evaluation of PDS on patients with at least 2 joint bleeds to diagnose early synovitis | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Suchitra S Acharya, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- New York Presbyterian Hospital/Hospital for Special Surgery, New York, New York, United States